CLINICAL TRIAL: NCT03961412
Title: Evaluation of A Family-based Intervention to Improve Pap Test Screening Among Under-screened Chinese American Immigrant Women
Brief Title: A Family-based Intervention to Improve Pap Test Screening Among Under-screened Chinese American Immigrant Women
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nevada, Reno (Other)
Responsible Party: Principal Investigator, Wei-Chen Tung, Associate Professor, PhD, RN, FAAN, San Jose State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 1440348-1
Record Dates: First submitted 2019-05-17; First posted 2019-05-23 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Cervical Cancer; Healthy Women
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- family-based intervention + education materials (Experimental): The participants will identify their accompanying influential person (e.g., spouse, partners, parents, children, friends) with whom they will be attending the 1.5-2 hour face-to-face education session on cervical cancer and screening. Their accompanying influential person is eligible if they are (a) aged 18 or older and (b) willing to participate in the study.
  Interventions: Behavioral: family-based intervention
- women only intervention + education materials (Active Comparator): Only the participants will attend the 1.5-2 hour face-to-face intervention on cervical cancer and screening.
  Interventions: Behavioral: Participant only intervention

INTERVENTIONS:
Behavioral: family-based intervention — The participants will identify their accompanying influential person(s) (e.g., spouse, partners, parents, children, friends) with whom they will be attending the 1.5-2 hour face-to-face education session on cervical cancer and screening. At the end of the intervention, time will be allowed for questions, as well as distributing fridge magnets and a pamphlet. Fridge magnets contain Pap test guidelines and availability of local clinics. The pamphlet covers the following topics: (a) information about female anatomy and cervical cancer, (b) risk factors for cervical cancer, (c) facts of cervical cancer incidence and mortality, and screening rates among American women, (d) methods to reduce cervical cancer (e.g., HPV vaccination), (e) Pap test procedure, (f) Pap test guidelines, and (g) availability of clinics and cost of Pap test. The participants will be encouraged to spread the message to family members and friends.
  Arms: family-based intervention + education materials
Behavioral: Participant only intervention — Only participant will attend the 1.5-2 hour face-to-face education session on cervical cancer and screening. At the end of the intervention, time will be allowed for questions, as well as distributing fridge magnets and a pamphlet. Fridge magnets contain Pap test guidelines and availability of local clinics. The pamphlet covers the following topics: (a) information about female anatomy and cervical cancer, (b) risk factors for cervical cancer, (c) facts of cervical cancer incidence and mortality, and screening rates among American women, (d) methods to reduce cervical cancer (e.g., HPV vaccination), (e) Pap test procedure, (f) Pap test guidelines, and (g) availability of clinics and cost of Pap test. The participants will be encouraged to spread the message to family members and friends.
  Arms: women only intervention + education materials

SUMMARY:
The purpose of this study is to find out the impact of the involvement of an influential person(s) (e.g., spouse, partners, parents, children, friends) on Pap test screening intention and behaviors, Pap test self-efficacy, and perceived benefits and barriers to Pap test screening among Chinese American immigrant women. These data specific to the impact of the involvement of an influential person on Pap test screening could be used to develop successful cancer prevention programs that target the specific needs of Chinese populations.

DETAILED DESCRIPTION:
The importance of the support from family, spouse, friends, or significant others has been noted among Chinese American immigrant women (CAIW), but little attention has been paid to the effects of family-based (FB) interventions, especially for cervical cancer screening. Understanding the role of CAIW's family in promoting Pap screening and other influences can lead to the creation of more culturally appropriate screening interventions. The objective of this study is to test the effects of a FB intervention on Pap test intention and behaviors, Pap test self-efficacy, and perceived benefits and barriers to Pap tests among under-screened CAIW aged 21-65. This pilot test of the FB intervention will be conducted using a randomized controlled design with two groups only, experimental and control groups. Interventions will be delivered by bilingual and bicultural CAIW trained facilitators. Post-test and follow-up telephone surveys will be conducted at 2 weeks and 6 months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* a first-generation Chinese American
* no previous cervical cancer screening within the past 3 years
* no total hysterectomy
* no history of cervical cancer
* able to read English, Simple Chinese, or Traditional Chinese.

Exclusion Criteria:

* Not a Chinese American immigrant
* Had total hysterectomy
* Had history of cervical cancer
* Not able to read English or Chinese

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 224 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change in Receiving a Pap Test | 2 weeks after intervention
  Change from baseline in use of a Pap test 2 weeks after intervention
Change in Receiving a Pap Test | 6 months after intervention
  Change from baseline in use of a Pap test 6 months after intervention
Change in Intention to Receive a Pap Test | 2 weeks after intervention
  Change from baseline in intention to receive a Pap test 2 weeks after intervention
Change in Intention to Receive a Pap Test | 6 months after intervention
  Change from baseline in intention to receive a Pap test 6 months after intervention

IPD SHARING:
Plan to Share IPD: No